CLINICAL TRIAL: NCT02250092
Title: Synergistic Effect of Combined Transcranial Direct Current Stimulation/Constraint Induced Movement Therapy in Children With Hemiparesis
Brief Title: Brain Stimulation and Hand Training in Children With Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Cerebral Palsy International Research Foundation (Other); Foundation for Physical Therapy, Inc. (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1408M53169
Record Dates: First submitted 2014-09-18; First posted 2014-09-26 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Pediatric Hemiparesis
Keywords: Cerebral Palsy; Hemiparesis; Stroke; Non-Invasive Brain Stimulation; Transcranial Direct Current Stimulation; Constraint-Induced Movement Therapy; Diffusion Tensor Imaging; Congenital Hemiparesis; Bimanual Therapy
MeSH Terms: conditions — Cerebral Palsy; Paresis; Stroke | interventions — Transcranial Direct Current Stimulation; Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- tDCS/CIMT (Active Comparator): Intervention Group will receive 20 minutes of 1.0 mA tDCS to the contralesional hemisphere concurrent with CIMT.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- tDCS sham/CIMT (Placebo Comparator): Placebo Group will receive 20 minutes of sham 1.0 mA tDCS to the contralesional hemisphere concurrent with CIMT.
  Interventions: Device: Placebo Comparator

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — 10 tDCS/CIMT Sessions
  Other Names: tDCS; Brain Stimulation
  Arms: tDCS/CIMT
Device: Placebo Comparator
  Arms: tDCS sham/CIMT

SUMMARY:
Hemiparetic cerebral palsy influences motor function in children during development and throughout their lifetime. The deficits one sees are the result both of the congenitally induced brain lesion and the subsequent plasticity that can impair function of the surviving neurons in the damaged brain.

Many current treatments have limited influence on children's neurorecovery. Constraint-induced movement therapy (CIMT) involving constraining the unaffected limb to encourage use of the affected limb has shown promise, yet with new technology revealing the potential to directly influence the brain, there is an urgent need to study the synergy of combined techniques.

Non-invasive brain stimulation (NIBS) as a direct neuromodulatory intervention has the potential to act synergistically with CIMT to influence neurorecovery.

Combining behavioral therapies, constraint-induced movement therapy (CIMT), with a novel form of neuromodulation, transcranial direct current stimulation (tDCS), we investigated the influence of this intervention on improved motor outcomes in children with cerebral palsy. The study hypotheses surround the safety, feasibility and efficacy of combined CIMT and tDCS wherein those children who receive the combined intervention will reveal no major adverse events, yet improved hand function and cortical excitability.

To Note: In addition to the combination of NIBS with CIMT, we also investigated the combination of NIBS with another form of motor intervention, bimanual, or two-handed, training. During bimanual training, children engage both hands in movements. The goal of bimanual training is to teach children how to most effectively use their hands cooperatively. During bimanual training, children play with games and toys that require the use of both hands. Children also practice activities of daily living that require the use of both hands, such as putting hair in a ponytail, tying shoes, and buttoning clothing. N=8 for this pilot study and no randomization. (Burke Medical Research Institute partnered with Columbia University and did a parallel pilot study. N=8 (PIs Friel and Gordon; Protocol BRC449)

DETAILED DESCRIPTION:
We use single-pulse transcranial magnetic stimulation (TMS) to measure the location and strength of brain connections that control hand movements.

ELIGIBILITY:
Inclusion Criteria:

1. Hemispheric Stroke or Periventricular Leukomalacia confirmed by most recent MRI or CT radiologic report with resultant congenital hemiparesis
2. ≥ 10 degrees of active motion at the metacarpophalangeal joint
3. Receptive language function to follow two-step commands as evidenced by performance on TOKEN test of intelligence
4. No evidence of seizure activity within the last 2 years
5. Presence of a motor evoked potential from at least the contralesional hemisphere if not both hemispheres
6. Ages 8-21 years
7. Able to give informed assent along with the informed consent of the legal guardian
8. Children who have had surgeries, which may influence motor function eg- tendon transfer, will be included, yet surgical history will be documented and included in any publication within a participant characteristics table.

Exclusion Criteria:

1. Metabolic Disorders
2. Neoplasm
3. Epilepsy
4. Disorders of Cellular Migration and Proliferation
5. Acquired Traumatic Brain Injury
6. Pregnancy
7. Indwelling metal or incompatible medical devices
8. Evidence of skin disease or skin abnormalities
9. Botulinum toxin or Phenol block within [six-months] preceding the study

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette T Gillick, PhD, MSPT, PT, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota

REFERENCES:
- [Background] Gillick B, Menk J, Mueller B, Meekins G, Krach LE, Feyma T, Rudser K. Synergistic effect of combined transcranial direct current stimulation/constraint-induced movement therapy in children and young adults with hemiparesis: study protocol. BMC Pediatr. 2015 Nov 12;15:178. doi: 10.1186/s12887-015-0498-1. PMID 26558386
- [Derived] Lixandrao MC, Stinear JW, Rich T, Chen CY, Feyma T, Meekins GD, Gillick BT. EMG breakthrough during cortical silent period in congenital hemiparesis: a descriptive case series. Braz J Phys Ther. 2020 Jan-Feb;24(1):20-29. doi: 10.1016/j.bjpt.2018.11.002. Epub 2018 Nov 22. PMID 30471965

RESULTS

PARTICIPANT FLOW:
Groups:
- tDCS Sham/CIMT: Placebo Group will receive 20 minutes of sham 1.0 mA tDCS to the contralesional hemisphere concurrent with CIMT.
  Placebo Comparator
Period: Overall Study
Arm/Group | tDCS/CIMT | tDCS Sham/CIMT
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | tDCS/CIMT | tDCS Sham/CIMT | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 8 | 18
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 12.33 (3.08) | 13.17 (5.08) | 12.7 (4.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 10 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 0 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Assisting Hand Assessment (AHA)
Description: Participants were videotaped while performing a bimanual age-appropriate activity. Investigators scored this performance using the Assessment of Assisting Hand (AHA) inventory. The AHA consists of 22 items, each scored on a 4-point scale. Raw scores are a sum of the 22 item scores, ranging from 22-88. Computer software logarithmically transforms ordinal raw scores into a final score. Final scores are reported on a logit-based AHA-unit scale and range from 0 to 100, with higher scores indicating greater ability. Outcome is reported as the change from baseline to 2 weeks and change from baseline to 6 months.
Time Frame: 2 weeks, 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | tDCS/CIMT | tDCS Sham/CIMT
Number analyzed (Participants) | 10 | 10
score on a scale
  2 weeks | 6.4 [3.4 to 9.4] | 8 [5.66 to 10.34]
  6 months | 5.5 [3.23 to 7.77] | 7.6 [3.92 to 11.28]

2. Secondary Outcome: Change in Canadian Occupational Performance Measurement (COPM)
Description: The COPM is clinician-administered semi-structured interview measuring the participant's perception of satisfaction and performance of personally set goals. There are 3 categories (Self-Care, Productivity, and Leisure) each containing 3 subcategories each for a total of 9 items, which are rated on an ordinal scale from 1 (minimum importance) to 10 (maximum importance). Each of the child's goals are given a satisfaction and performance rating. The average of the satisfaction ratings across all goals is reported as the "average satisfaction score", ranging from 1 to 10, with higher scores indicating a better outcome. Outcome is reported as the change from baseline to 2 weeks and change from baseline to 6 months.
Time Frame: 2 weeks, 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | tDCS/CIMT | tDCS Sham/CIMT
Number analyzed (Participants) | 10 | 10
score on a scale
  2 weeks | 2.14 [1.23 to 3.05] | 1.8 [1.27 to 2.33]
  6 months | 2.94 [2.04 to 3.84] | 3.22 [2.57 to 3.87]

3. Other Pre Specified Outcome: Change in Subject Symptom Assessment (SSA) From 2 Weeks to 6 Months
Description: The Subject Symptom Assessment (SSA) is a questionnaire of common side effects reported in the literature that is asked of the child undergoing non-invasive brain stimulation. This measure asks the child to rate if the symptom is present (yes or no) and if it is present, rate the severity using a 1 to 4 scale (1 indicates absent, 2=mild, 3=moderate, 4=severe). Lower values are better as they represent absent or mild symptoms. Outcome is reported as the change in symptom severity from 2 weeks of treatment to 6 months of treatment. This measure is not collected at baseline.
Time Frame: 2 weeks, 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | tDCS/CIMT | tDCS Sham/CIMT
Number analyzed (Participants) | 10 | 10
score on a scale | 1.7 [0.5 to 2.9] | 1.76 [0.96 to 2.56]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | tDCS/CIMT | tDCS Sham/CIMT
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS/CIMT (N=10) | tDCS Sham/CIMT (N=10)
Headache (General disorders) | 4 (9) | 1 (1)
Unusual Feelings on the Skin of the Head (General disorders) | 2 (5) | 1 (1)
Itchiness (General disorders) | 1 (5) | 3 (6)
Unusual Feelings or Emotions (General disorders) | 1 (2) | 0 (0)
Dizziness (General disorders) | 0 (0) | 3 (3)
Nausea (General disorders) | 0 (0) | 1 (1)
Tingling (General disorders) | 2 (10) | 2 (2)
Difficulty Paying Attention (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT02250092/Prot_SAP_000.pdf